CLINICAL TRIAL: NCT04096352
Title: Virtual Reality in Teachers' Vocal Motor Behavior Acquisition (VirtuVox): Randomized Controlled Trial
Brief Title: Virtual Reality in Teachers' Vocal Motor Behavior Acquisition (VirtuVox)
Acronym: VirtuVox
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Collaborators: Universite du Quebec en Outaouais (Other)
Responsible Party: Principal Investigator, Remacle Angélique, Principal Investigator, University of Liege
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: VirtuVox2
Record Dates: First submitted 2019-09-06; First posted 2019-09-19 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Voice Disorders; Virtual Reality Therapy
Keywords: Speech Therapy; Virtual Reality; Teacher's voice; Background Noise; School Teachers
MeSH Terms: conditions — Voice Disorders; Communication Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Indirect+Direct method (Experimental): Indirect method: one session of information on voice function and voice hygiene.
  Direct method: three sessions of voice training using virtual reality simulations over a course of 3 weeks.
  Interventions: Behavioral: Direct Method; Behavioral: Indirect Method
- Indirect method (Active Comparator): Indirect method: one session of information on voice function and voice hygiene.
  Interventions: Behavioral: Indirect Method

INTERVENTIONS:
Behavioral: Direct Method — Learning effective vocal skills using speech therapy exercises and virtual reality simulations.
  Arms: Indirect+Direct method
Behavioral: Indirect Method — Information on voice function and voice hygiene.

SUMMARY:
Scientific literature supports that teachers are at greater risk for voice disorders than the general population. In the classroom, the teacher's voice represents the main communication tool. Optimal voice use is indispensable to ensure effective teaching and preserve the teacher's vocal health.

This project investigates how virtual reality (VR) facilitates the learning of effective vocal skills and their application in real-world contexts. Based on acoustic analyses and self-assessment scales, the investigators compare 100 future teachers randomly assigned in two groups. The experimental group (n=50) receives a voice training by VR simulations and voice information. The control group (n=50) only receives voice information.

DETAILED DESCRIPTION:
Experimental group participants receive direct method (three 1-hour sessions of voice training by virtual reality simulations over a course of 3 weeks) and indirect method (one 1-hour session of information on voice function and voice hygiene). Control group participants receive indirect method (one 1-hour session of information on voice function and voice hygiene).

ELIGIBILITY:
Inclusion Criteria:

* future teacher having completed at least one internship as a schoolteacher
* speaking French fluently

Exclusion Criteria:

* hearing impairment
* voice pathology at the time of the study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2019-09-29 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
Self-perceived voice changes between the baseline and the end of the intervention | 3 weeks
  Self-assessment of perceived vocal effort using the Adapted BORG Category Ratio (CR-10) physical exertion scale. On the scale, verbal expressions regarding vocal effort are anchored to the correct positions on a logarithmic ratio scale from zero (No vocal effort at all) to 10 (Maximum vocal effort), according to their quantitative meaning.
Voice frequency changes between the baseline and the end of the intervention | 3 weeks
  Acoustic measurements of participants' voice frequency (in hertz) when speaking with and without background noise.
Voice intensity changes between the baseline and the end of the intervention | 3 weeks
  Acoustic measurements of participants' voice intensity (in dB) when speaking with and without background noise.
Voice spectrum changes between the baseline and the end of the intervention | 3 weeks
  Acoustic measurements of participants' voice spectrum (in Hertz) when speaking with and without background noise.
Speech rate changes between the baseline and the end of the intervention | 3 weeks
  Measurements of participants' speech rate (in syllables per second) when speaking with and without background noise.

CONTACTS AND LOCATIONS:
Overall Officials: Angélique Remacle, Ph.D., Principal Investigator — University of Liege
Locations (1):
- Université de Liège, Liège, Wallonia, Belgium